CLINICAL TRIAL: NCT00909207
Title: Refinement of the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Via Cognitive Interviewing and Usability Testing
Brief Title: Patient-Reported Outcomes Version of Common Terminology Criteria (CTCPRO) Cognitive Debriefing
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2009-0182
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Cancers; Hematologic Diseases; Solid Tumors
Keywords: Advanced Cancers; Hematologic Disorders; Solid Tumors; Cognitive Interview; Patient-Reported Outcomes; PRO; Common Terminology Criteria for Adverse Events; CTCAE; PRO-CTCAE; Cancer Symptoms; Interview
MeSH Terms: conditions — Hematologic Diseases | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interview: Review list of 25 cancer symptoms, 20-30 minute audio-taped personal interview and 15-20 minute questionnaire.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Review list of 25 cancer symptoms, 20-30 minute audio-taped personal interview and 15-20 minute questionnaire.

SUMMARY:
The scientific aim of this study is to evaluate patient comprehension of the 77 newly developed items as well as the extent to which the items correspond to the concepts of interest for each patient reported outcome (PRO).

A secondary aim of this study is to evaluate the usability of the technology interface for collecting the PRO data of the PRO-CTCAE system once it has been built to accommodate the learning garnered during the cognitive interviews.

DETAILED DESCRIPTION:
Screening:

The study staff will talk to your doctor or nurse, and/or look at your medical record, to see if you are currently receiving treatment. The study staff will also look at your medical record to see if you have any future clinic visits at M. D. Anderson. This is the first step of "screening" to help the researchers decide if you are eligible to take part in this study.

If you are found to be possibly eligible to take part in this study based on the first step of screening, the second step of screening will occur:

At your clinic visit, the study staff will talk to you about this study. You will be asked questions about school, which should take about 2 minutes.

Study Visit If you are found to be eligible and you agree to take part in this study, you will look at a list of 34 cancer symptoms if you are a male or a list of 36 cancer symptoms if you are a female. You will fill out a questionnaire that asks you to mark each symptom that you may be experiencing at this time, and other information about the symptoms such as how often they occur.

After you complete the questionnaire, you will be interviewed by the study staff about how you answered some of the questions. For example, you will be asked if the words describing the symptoms were easy to understand or if other words may be more clear.

There are no right or wrong answers to any part of this study. Researchers are interested in your thoughts about the words.

Filling out the questionnaire will take about 10-15 minutes. The interview will take about 20-30 minutes.

Study Data:

The interview will be audio-recorded. Only the study staff will hear the recording. The recording will be saved on a password-protected computer that can only be accessed by the study staff.

Your responses will be coded without using your name or other personal identifying information. Only the study staff will have access to the code numbers and be able to identify you.

Your responses will not be shared with your doctor without your consent.

In some of the questions, you will be asked about your feelings (for example, whether you feel unhappy or anxious). If your responses show that you may be having emotional difficulties, you will be given a list of community agencies that provide services for emotional issues. You may also speak to your doctor about your feelings.

Length of Study:

After the study visit, your active participation will be over. In some cases, the study staff may call you to ask that you clarify some of your answers. Your medical record may also be checked to confirm the cancer diagnosis and your treatments.

This is an investigational study. Up to 100 patients will take part in this study. Up to 20 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be aged 18 and over
2. Able to read and understand English
3. Patients with a high school education or less
4. Patients who are undergoing chemotherapy or radiotherapy with curative or palliative intent.
5. Patient is able to provide informed consent.
6. All types of cancer diagnosis

Exclusion Criteria:

1) Significant cognitive impairment as determined by research staff's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals, age 18 years or older, receiving chemotherapy and/or radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Comprehension of Patient Reported Outcome (PRO) Criteria | 1 day
  The primary assessment tool will be the cognitive interview protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Tito Mendoza, PhD, MS, MED, Study Chair — UT MD Anderson Cancer Center
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.clinicaltrials.org